CLINICAL TRIAL: NCT07389096
Title: Opioid-Free Anesthesia Versus Opioid Based Anesthesia For Adolescent Idiopathic Scoliosis A Prospective Randomized Double-Blind Controlled Trial
Brief Title: Opioid-Free Anesthesia Versus Opioid Based Anesthesia For Adolescent Idiopathic Scoliosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nashwa Ahmed (Other)
Responsible Party: Sponsor-Investigator, Nashwa Ahmed, , Lecturer of Anaesthesia and Surgical Intensive Care, Faculty of Medicine, Port Said University, Egypt, Port Said University hospital
Organization: Port Said University hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB00012098- Serial0307600
Record Dates: First submitted 2025-12-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Opioid Free Anesthesia
MeSH Terms: interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group OFA (Opioid-Free Anesthesia): (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- Group OBA (Opioid-Based Anesthesia) (Active Comparator)
  Interventions: Drug: Fentanyl (IV)

INTERVENTIONS:
Drug: Dexmedetomidine — patients will Receive dexmedetomidine with a loading dose of 1 μg/kg followed by a maintenance infusion of 0.5 μg/kg/h.
  Arms: Group OFA (Opioid-Free Anesthesia):
Drug: Fentanyl (IV) — patients will Receive fentanyl with a loading dose of 1 μg/kg followed by a maintenance infusion of 0.5 μg/kg/h.
  Arms: Group OBA (Opioid-Based Anesthesia)

SUMMARY:
Opioid-free anesthesia (OFA) is a multimodal analgesic approach designed to eliminate the intraoperative use of systemic, neuraxial, or intracavitary opioids. This technique employs a combination of antinociceptive agents targeting various pathways within the central and peripheral nervous systems to achieve effective analgesia.

Dexmedetomidine (DEX), a highly selective α2-adrenoreceptor agonist, is a centrally acting non-opioid agent increasingly utilized in clinical practice for its antinociceptive and anxiolytic properties. Only a few prospective randomized controlled trials have specifically examined the postoperative analgesic efficacy of intraoperative dexmedetomidine infusion in patients undergoing spinal surgery, with limited data focusing on this as a primary endpoint. Importantly, no clinical studies have investigated its analgesic impact in patients undergoing spinal surgery under general anesthesia.

DETAILED DESCRIPTION:
Reducing perioperative opioid exposure presents a critical opportunity for anesthesiologists, surgeons, and institutions to minimize patient harm and improve recovery outcomes. Opioid-free anesthesia (OFA) has emerged as a promising approach to address this need. Opioid-free anesthesia is defined as an anesthetic technique that excludes intraoperative opioid administration through all routes including systemic, neuraxial, and local tissue infiltration relying instead on multimodal non-opioid strategies to achieve effective analgesia. (5) Aim This study explores the intraoperative and postoperative application of dexmedetomidine (DEX) as an opioid-free anesthetic strategy to improve perioperative outcomes in patients undergoing scoliosis surgery under general anesthesia.

Hypothesis:

Continuous infusion of Dexmedetomidine at 0.5 μg/kg/h, following an initial loading dose of 1 μg/kg, yields more effective than standard approaches.

Outcomes This prospective randomized controlled study investigates the intraoperative and postoperative efficacy of dexmedetomidine (DEX) infusion in patients undergoing scoliosis surgery. The primary outcome is intraoperative analgesic effectiveness, while secondary outcomes include the incidence of perioperative complications, the requirement for rescue fentanyl, and surgeon satisfaction.

Thirty patients will be prospectively enrolled and randomly allocated into two parallel groups:

* Group OFA (Opioid-Free Anesthesia): patients will Receive dexmedetomidine with a loading dose of 1 μg/kg followed by a maintenance infusion of 0.5 μg/kg/h.
* Group OBA (Opioid-Based Anesthesia): patients will Receive fentanyl with a loading dose of 1 μg/kg followed by a maintenance infusion of 0.5 μg/kg/h.

Methods Ethics committee approval will be obtained, and written informed consent will be secured from the parents of each pediatric participant.

We will conduct a prospective, randomized study involving 30 pediatric patients aged 8 to 18 years, diagnosed with idiopathic scoliosis and will be scheduled for surgical correction. Patients will be randomly assigned into two equal groups.

Anesthetic technique Preoperative Routine Preoperative Investigations

The standard preoperative workup included:

* Complete Blood Count (CBC)
* Electrocardiogram (ECG) and Echocardiography
* Coagulation Profile
* Blood Urea Nitrogen (BUN) and Serum Electrolytes
* Blood Crossmatch Additional Investigations
* Plain Chest Radiography
* Arterial Blood Gas (ABG) Analysis
* Pulmonary Function Tests (PFTs), routinely performed to detect restrictive lung defects During the evening preceding surgery, patients will be educated on the use of a five-point visual analog pain scale, illustrated by a series of facial expressions. This scale is designed to facilitate self-assessment, with 1 denoting no pain and 5 indicating the worst imaginable pain. (2) Intraoperative Upon arrival to the operating room, standard monitoring is initiated in accordance with American Society of Anesthesiologists (ASA) guidelines. This includes continuous five-lead electrocardiography, non-invasive blood pressure, pulse oximetry, capnography, core temperature monitoring, and urine output measurement.

Patients will receive intravenous hydration with 0.9% normal saline at 5-6 mL/kg to maintain adequate systolic blood pressure. No premedication is administered. Hypothermia prevention will be achieved using forced warm air devices.

Antibiotic prophylaxis is administered appropriately within 30 minutes prior to skin incision.

Induction of anesthesia will be achieved with an intravenous bolus of propofol at 2 mg/kg, followed by atracurium at 0.5 mg/kg to facilitate orotracheal intubation. No additional neuromuscular blocking agents are administered during the procedure.

Mechanical ventilation will be maintained using a 1:1 oxygen-to-air mixture (FiO₂ 0.5), with a tidal volume of 6-8 mL/kg and a respiratory rate is adjusted between 8 and 14 breaths per minute to maintain end-tidal CO₂ levels within the range of 30-35 mmHg

Following induction, all patients will receive the following intravenous infusions:

1. Propofol is administered at 50-150 μg/kg/min, will be titrated to maintain mean arterial pressure (MAP) within ±20% of baseline values.
2. Continuous propofol infusion is similarly adjusted across both study groups to ensure adequate anesthetic depth. Inadequate anesthesia is defined as a heart rate exceeding pre-induction values by more than 15% and/or systolic arterial pressure exceeding baseline by more than 20%, persisting for at least one minute in the absence of hypovolemia or low hematocrit.
3. A total of 4 g of intravenous magnesium sulfate will be administered intraoperatively.
4. Tranexamic acid will be administered as a loading dose of 15 mg/kg, followed by a continuous infusion at 5 mg/kg/hr, continued until completion of surgical hemostasis.

In Group D (Dexmedetomidine) Patients will be administered a loading dose of dexmedetomidine at 1 μg/kg over 10 minutes, followed by a continuous infusion at 0.5 μg/kg/hr.

For consistency in preparation, 200 μg of dexmedetomidine [Precedex®, Pfizer] is diluted with normal saline in a 50 mL syringe, resulting in a final concentration of 4 μg/mL.

In Group F (Fentanyl):

Patients will receive opioid-based anesthesia (OBA) consisting of a fentanyl loading dose of 1 μg/kg, followed by a maintenance infusion at 0.5 μg/kg/hr.

An additional large-bore 16-gauge intravenous cannula will be placed in the contralateral hand to serve as a transfusion access line.

Ringer's lactate is administered via an intravenous fluid warmer at a rate of 10 mL/kg/hr, with blood products will be supplemented as clinically indicated.

A Foley catheter is inserted in all patients and will be connected to a urine collection bag for continuous monitoring of urinary output.

Following catheterization, patients are carefully positioned prone, with meticulous attention to the eyes, airway, and pressure points, all of which are assessed, supported, and protected to prevent positioning related complications.

Following placement of the spinal rod instrumentation, the orthopedic surgeon requests a wake-up test, a procedure is considered the gold standard for intraoperative neurological assessment during scoliosis correction surgery. (6) At this point, dexmedetomidine and fentanyl infusions will be discontinued.

After the patient has reached an appropriate level of consciousness for testing. The patient is instructed to grip his hands to assess responsiveness, followed by a command to move his feet. Both tasks are successfully performed without any adverse events, such as excessive movement, accidental extubation, or risk of falling.

Upon completion of the test, anesthesia will be re-established with an intravenous bolus of propofol (2 mg/kg) and atracurium (0.5 mg/kg). The depth of anesthesia will be maintained at the same level as prior to the wake-up test, and the surgical procedure proceeded without complications.

To initiate emergence from anesthesia, the infusion rate of the maintenance anesthetic agent is reduced to 50% at the onset of surgical closure and is discontinued once the patient is repositioned supine. All patients will receive ondansetron (0.1 mg/kg) for antiemetic prophylaxis and paracetamol (15 mg/kg) for analgesia.

Neuromuscular reversal will be achieved using a standard protocol, neostigmine (0.05 mg/kg) is combined with glycopyrrolate (0.01 mg/kg), will be administered upon confirmation of a train-of-four (TOF) count of 4 and a TOF ratio exceeding 80%. Extubation is performed in supine position, contingent upon clinical indicators of full recovery including adequate spontaneous respiration and responsiveness to verbal commands and a TOF ratio >0.9.

Postoperatively Patients will be transferred to either the high dependency unit (HDU) or the neurosurgical intensive care unit (NICU). All patients will receive intravenous paracetamol (15 mg/kg every 6 hours) for 48 hours to maintain analgesia.

Measurements Intraoperative Haemodynamics Heart rate (HR) and blood pressure (BP) will be continuously monitored using non-invasive techniques at 30-minute intervals throughout the procedure. Specific hemodynamic data points will be recorded at baseline, during skin incision, at 30 minutes post-incision, during skin closure, and at extubation, will be documented in the anesthesia follow-up records.

In all cases, increases in mean arterial pressure (MAP >100 mmHg) or heart rate exceeding 15% above baseline are managed with incremental boluses of propofol, up to 50 mg per dose, is tailored to the patient's response.

Assessment of Intraoperative Blood Loss The visual estimation method remains the most employed technique for assessing intraoperative blood loss in clinical practice. This approach involves evaluating the volume of blood collected in suction canisters, the degree of saturation of surgical gauze, and the visible blood within the operative field.(7) Surgeon Satisfaction Assessment (8)

Surgeon satisfaction will be evaluated in both groups using Likert scale, with scores ranging from 1 to 5, corresponding to the following levels:

1 = Very Bad, 2 = Bad, 3 = Average, 4 = Good, and 5 = Excellent . Satisfaction ratings are recorded postoperatively to assess the perceived quality of surgical conditions and overall intraoperative experience.

Quality of surgical field (9)

The quality of surgical field will be evaluated every 30 min using the surgical field rating (SFR) scale of six points proposed by Fromme et al.:

5- massive uncontrollable bleeding 4- heavy but controllable bleeding that significantly interfered with dissection 3- moderate bleeding that moderately compromised surgical dissection 2-moderate bleeding a nuisance but without interference with accurate dissection

1- bleeding, so mild it is not even a surgical nuisance 0- no bleeding and virtually bloodless field.

Surgical field was graded as good, fair, and poor as:

good - SFR scale 0 or 1 fair - SFR scale 2 or 3 poor - SFR scale 4 or 5 Postoperative Recovery Assessment Post-anesthesia recovery is evaluated using the Post Anesthesia Recovery Score (PARS), alongside measurement of immediate recovery time, defined as the interval from discontinuation of dexmedetomidine or fentanyl infusion to the patient's response to verbal command by opening the eyes. Assessments are conducted at 5-minute intervals starting from the cessation of the anesthetic infusion. (2) Pain Assessment and Analgesic Intervention (3)

Postoperative pain will be assessed at 2, 6, 12, 24 hours using the Numerical Rating Scale (NRS). Pain intensity is classified as follows:

* Mild: NRS 1-3
* Moderate: NRS 4-6
* Severe: NRS 7-10 Intravenous fentanyl (1 µg/kg) is administered as rescue analgesia when the NRS score exceeded 4. The pain free interval is defined as the duration between cessation of the study anesthetic agent and the first administration of rescue analgesia.

Postoperative Complications

Patients are monitored for the following adverse events:

* Nausea and vomiting
* Shivering
* Pruritus
* Respiratory desaturation, defined as peripheral oxygen saturation (SpO₂) < 92%

ELIGIBILITY:
Inclusion Criteria:Patients younger than 18 years of age, classified as American Society of Anesthesiologists (ASA) Physical Status I or II, and will be scheduled for surgical correction of adolescent idiopathic scoliosis.

-

Exclusion Criteria:• Refusal to participate in the study or to allow use of personal data

* Non-idiopathic scoliosis
* Contraindications to commonly used perioperative medications
* ASA Physical Status ≥ III
* Presence of neuromuscular disorders or severe cardiac dysfunction
* Requirement for postoperative mechanical ventilation
* Regular use of analgesics or opioids
* History of allergy to opioids or dexmedetomidine
* Diagnosed mental disorders
* Severe hepatic or renal dysfunction
* Coagulopathy or significant pulmonary disease
* Preoperative or postoperative neurological deficits
* Occurrence of serious arrhythmia, hypotension, or bradycardia necessitating discontinuation of dexmedetomidine infusion

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
intraoperative analgesic effectiveness, Measured by Heart Rate | 2 hours
  Changes in heart rate recorded at predefined intraoperative intervals to assess physiological response to analgesia.
intraoperative analgesic effectiveness, Measured by blood pressure | 2 hours
  Changes in blood pressure recorded at predefined intraoperative intervals.

SECONDARY OUTCOMES:
the requirement for rescue fentanyl | 24 hour
  Postoperative pain was assessed at 2, 6, 12, 24 hours using the Numerical Rating Scale (NRS).
surgeon satisfaction | 2 hours
  using Likert scale, with scores ranging from 1 to 5,
Assessment of Intraoperative Blood Loss | 2 hours
  evaluating the volume of blood collected in suction canisters, the degree of saturation of surgical gauze, and the visible blood within the operative field
hemodynamics | 2 hours
  Heart rate (HR) and blood pressure (BP) were continuously monitored using non-invasive techniques at 30-minute intervals throughout the procedure.
Quality of surgical field | 2 hours
  the surgical field rating (SFR) scale of six points proposed by Fromme et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Port said university, Port Said, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aujla KS, Kaur M, Gupta R, Singh S, Bhanupreet, Tavleen. A study to compare the quality of surgical field using total intravenous anesthesia (with propofol) versus inhalational anesthesia (with isoflurane) for functional endoscopic sinus surgeries. Anesth Essays Res 2017; 11:606-10. DOI: 10.4103/0259-1162.206858
- [Result] Ghorbani J, Arastou S, Naeini A, Raad N, Galougahi M, Jahangirifard A, Dilmaghani N. Comparing the Effect of Oral Clonidine and Tranexamic Acid on Bleeding and Surgical Field Quality during Functional Endoscopic Sinus Surgery. Iranian Journal of Otorhinolaryngology 2018; 30(5):255-60
- [Result] Lin Y, Yu C, Xian G. Calculation methods for intraoperative blood loss: a literature review. BMC Surgery 2024; 24:394 doi.org/10.1186/s12893-024-02699-3
- [Result] Pipat Saeyup, Chanon Thanaboriboon. Anesthetic Management and Role of Dexmedetomidine During Intraoperative Wake Up Test in Juvenile Idiopathic Scoliosis Correction Surgery: A Case Report. International Journal of Anesthesia and Clinical Medicine. 2019; 7(1): 27-30 Doi: 10.11648/j.ijacm.20190701.15
- [Result] Soffin E, Wetmore D, BeckmanJ, Sheha E, Vaishnav A, Albert T, Gang C, Qureshi S. Opioid-free anesthesia within an enhanced recovery after surgery pathway for minimally invasive lumbar spine surgery: a retrospective matched cohort study. Neurosurg Focus 2019;46(4): E8.DOI: 10.3171/2019.1. FOCUS18645
- [Result] 4- Çatalca, Sibel, Özmete, Özlem, Berk, Numan, Çivi, Soner, Durdağ, Emre, Incekaş, Caner, Özyilkan, Nesrin Bozdoğan. Does dexmedetomidine infusion reduce the postoperative analgesic need in lumbar disc surgery? Turkish Journal of Medical Sciences 2025;55: 470-481. doi.org/10.55730/1300-0144.5991
- [Result] 3- Rani US, Panda NB, Chauhan R, Mahajan S, Kaloria N, Tripathi M. Comparison of the effects of opioid free anesthesia (OFA) and opioid based anesthesia (OBA) on postoperative analgesia and intraoperative hemodynamics in patients undergoing spine surgery: A prospective randomized double blind controlled trial. Saudi J Anaesth 2024; 18:173 80. DOI: 10.4103/sja.sja_341_23
- [Result] 2- Moustafa A, Negmi H, Rabie M. The Combined effect of ketamine and remifentanil infusions as total intravenous anesthesia for scoliosis surgery in children. Middle East J Anaesthesiol 2008 ;19(5):1151-68.
- [Result] 1- Ferschl M, Shibata G, Wong J. New Surgical Approaches to Scoliosis Repair in Pediatric Patients Implications for Anesthetic Management. Current Anesthesiology Reports 2024; 14:475-83. doi.org/10.1007/s40140-024-00641-0